CLINICAL TRIAL: NCT01351298
Title: Intra-nasal Topical Local Anesthetic and Decongestant for Flexible Nasendoscopy in Children: a Randomised Double-blind Placebo Controlled Trial
Brief Title: Nasal Prep for Nasendoscopy in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's & Women's Health Centre of British Columbia (Other)
Responsible Party: Principal Investigator, Neil Chadha, Clinical Assistant Professor, Children's & Women's Health Centre of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H11-00602
Record Dates: First submitted 2011-05-06; First posted 2011-05-10 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Flexible Nasendoscopy
MeSH Terms: interventions — xylometazoline; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Saline spray (Placebo Comparator)
  Interventions: Drug: Isotonic normal saline
- Decongestant (Experimental)
  Interventions: Drug: 0.05% xylometazoline hydrochloride
- Decongestant and local anesthetic (Experimental)
  Interventions: Drug: 0.05% xylometazoline hydrochloride with 1% lidocaine hydrochloride

INTERVENTIONS:
Drug: 0.05% xylometazoline hydrochloride with 1% lidocaine hydrochloride — Decongestant with local anesthetic
  Arms: Decongestant and local anesthetic
Drug: 0.05% xylometazoline hydrochloride — Decongestant
  Arms: Decongestant
Drug: Isotonic normal saline — Placebo
  Arms: Saline spray

SUMMARY:
Flexible nasendoscopy involves passing a soft, thin, endoscope through the nose. This diagnostic procedure is often essential for assessment of a child by an Otolaryngologist in outpatients. The purpose of this randomized controlled double-blind study is to determine whether there is a difference in the degree of discomfort experienced by children undergoing flexible nasendoscopy, after receiving one of three different intranasal sprays: (A) placebo (isotonic saline solution), (B) decongestant (0.05% xylometazoline hydrochloride), or (C) decongestant with local anesthetic (0.05% xylometazoline hydrochloride with 1% lidocaine hydrochloride).

Null hypothesis: There is no difference in the degree of reported discomfort experienced (using a validated pediatric pain score) by children undergoing flexible nasendoscopy, after receiving either intra-nasal topical placebo, decongestant, or decongestant with local anesthetic.

ELIGIBILITY:
Inclusion Criteria:

* Fully informed consent from parent/caregiver
* Children aged 3 to 12 years
* Children deemed to require flexible nasendoscopy as part of their assessment during a Pediatric Otolaryngology clinic visit

Exclusion Criteria:

* Children who have previously undergone this procedure
* Children with current upper respiratory tract infection
* Children with known allergy to any of the trial medications

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Pain score (self) | Immediately post-nasendoscopy - same day as administration of nasal prep agent (day 1)
  Self-reported Wong-Baker Faces Pain Score

SECONDARY OUTCOMES:
Pain score (proxy) | Immediately post-nasendoscopy- same day as administration of nasal prep agent (day 1)
  The caregiver-proxy Wong-Baker Faces Pain Score
Ease of nasendoscopy score | Immediately post-nasendoscopy- same day as administration of nasal prep agent (day 1)
  Visual analog scale endoscopist rating

CONTACTS AND LOCATIONS:
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Chadha NK, Lam GO, Ludemann JP, Kozak FK. Intranasal topical local anesthetic and decongestant for flexible nasendoscopy in children: a randomized, double-blind, placebo-controlled trial. JAMA Otolaryngol Head Neck Surg. 2013 Dec;139(12):1301-5. doi: 10.1001/jamaoto.2013.5297. PMID 24158493